CLINICAL TRIAL: NCT00859794
Title: An Examination of Cognitive and Sensorimotor Processes in Patients With Epilepsy Using Electrophysiology, Cortical Mapping, Electrical Brain Stimulation, and fMRI
Brief Title: An Examination of Cognitive and Sensorimotor Processes in Patients With Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-125
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; fMRI; Electrophysiology; Cortical Mapping; Neurosurgery
MeSH Terms: conditions — Epilepsy | interventions — Neuropsychological Tests; Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive and Behavioral Testing (Experimental): Participants will participate in cognitive tasks where brain recordings and task performance will be monitored and recorded.
  Interventions: Other: fMRI; Other: Neuropsychological Testing; Other: Additional electrode implantation; Other: Electrical brain stimulation

INTERVENTIONS:
Other: fMRI — Subjects will perform cognitive tasks during MRI scanning sessions to gather data about cognitive functions.
Other: Neuropsychological Testing — Subjects will have a neuropsych evaluation as part of their standard of care for surgery. The research team is asking the subject to release their neuropsychological evaluations for analysis.
Other: Additional electrode implantation — Subjects will typically have between 100-300 electrodes implanted as part of their surgery. Additional electrodes will be implanted that are able to record from smaller, more specific parts of the brain. This will allow for better understanding of how the brain is wired.
Other: Electrical brain stimulation — Intracranial or extracranial electrodes will be used to deliver electrical brain stimulation (amplitude 0.5-8.0mA) or sham stimulation of between 0.4 and 3000 milliseconds during cognitive task periods.

SUMMARY:
The overall goal of this project is to better understand the micro-physiology of human epilepsy and cognition using the intracranial electroencephalogram (iEEG), electrical brain stimulation, functional magnetic resonance imaging (fMRI), and histology.

DETAILED DESCRIPTION:
The overall goal of this project is to better understand the micro-physiology of human epilepsy and cognition using iEEG, electrical brain stimulation, fMRI, and histology.

Specific AIM 1: Mapping cognitive networks using intracranial electrodes, functional magnetic resonance imaging, and cognitive tasks. To identify brain areas and mechanisms involved in cognitive function we will ask participants to perform tasks while their brain activity is measured with intracranial electrodes or functional magnetic resonance imaging (fMRI).

Specific AIM 2: Using microelectrodes to better understand the mechanisms of seizure genesis/spread and human cognitive function. We will use microelectrodes to measure activity within single neurons, data that will allow us to tease apart incoming and outgoing activity to a brain area.

Specific AIM 3: Using macroscale measures of brain connectivity to map functional and epileptogenic brain areas. We will measure connectivity between macroscale brain regions via variety of techniques: diffusion tensor imaging (DTI), fMRI, cortico-cortical evoked potentials (CCEP), and intracranial electrophysiology. We believe that epileptogenic and functional regions will be mutually segregated by their connectivity patterns.

Specific AIM 4: Using EEG/iEEG source localization to better identify the sources of epileptiform activity. We will construct models of participants' heads via MRI and CT, which will potentially allow us to localize the neural generators of EEG and iEEG recordings.

Specific AIM 5: Investigating the effects of transcranial and direct electrical stimulation on cortical excitability and cognitive function. We will apply direct electrical brain stimulation to epileptogenic and functional brain regions and evaluate the effects of this stimulation on electrode recordings, CCEPs, and cognitive tasks. Electrical stimulation may be applied with consideration of endogenous cognitive biomarkers to probe and elucidate the function of these biomarkers as they relate to cognitive function.

Specific AIM 6: Studying local connectivity of epileptic brain tissue with histology. We will reserve a small portion of resected brain tissue from patients who have undergone surgical resection for histological analysis to better understand altered patterns of neural connectivity in epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are selected on the basis of intractability of their seizures to medical intervention by antiepileptic drugs and following a noninvasive workup that indicates the patient would be an excellent candidate for resective surgery.

Exclusion Criteria:

* Patient is under the age of 5

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2007-11; Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Decrease in seizure frequency after epilepsy surgical treatment | up to 4 weeks
  We are interested in identifying specific factors that predict the effects of epilepsy surgery on seizure control. We will start by assessing electrographic (seizure foci and spread), imaging (cortical volume, presence of structural pathology), and surgical (extent of surgical resection) factors.
Change in electrophysiological markers (local field potential power and phase) during cognitive tasks | up to 4 weeks
  We will compare brain recordings during distinct cognitive functional states, as defined by performance and participation in cognitive tasks (typically task vs resting state). Power and phase measures isolated from local field potentials in implanted electrodes will be assessed. Neuronal firing rates will also be assessed.
Change in memory performance | up to 4 weeks
  We will measure the change in memory performance in memory tasks (percent of items correctly recalled).
Change in decision-making performance | up to 4 weeks
  We will measure the change in performance (reaction time and accuracy) in decision-making tasks.
Change in sensory perception | up to 4 weeks
  We will measure the change in performance in auditory/visual perception tasks (percent of items correctly perceived).

CONTACTS AND LOCATIONS:
Overall Officials: Ashesh Mehta, M.D., Ph.D., Principal Investigator — Zucker School of Medicine at Hofstra/Northwell and Feinstein Institute for Medical Research
Locations (1):
- Comprehensive Epilepsy Care Center, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided